CLINICAL TRIAL: NCT02039726
Title: A Phase 3 Open-label Randomized Study of Quizartinib (AC220) Monotherapy Versus Salvage Chemotherapy in Subjects With Tyrosine Kinase 3 - Internal Tandem Duplication (FLT3-ITD) Positive Acute Myeloid Leukemia (AML) Refractory to or Relapsed After First-line Treatment With or Without Hematopoietic Stem Cell Transplantation (HSCT) Consolidation
Brief Title: (QuANTUM-R): An Open-label Study of Quizartinib Monotherapy vs. Salvage Chemotherapy in Acute Myeloid Leukemia (AML) Subjects Who Are FLT3-ITD Positive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC220-007; EudraCT Number 2013-004890-28 (Other: Universal Trial Number (UTN) U1111-1151-8078)
Record Dates: First submitted 2014-01-15; First posted 2014-01-20 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: AML
Keywords: Acute Myeloid Leukemia; AML; FMS-like tyrosine kinase 3; FLT3-ITD; Quizartinib; Leukemia; Tablets
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — quizartinib; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quizartinib (Experimental): Participants who were randomized to receive 20 or 30 mg quizartinib tablets administered orally once daily.
  Interventions: Drug: Quizartinib
- Salvage chemotherapy (Active Comparator): Participants who were randomized to receive salvage chemotherapy, such as low dose cytarabine (LoDAC); mitoxantrone, etoposide, and intermediate-dose cytarabine (MEC); or fludarabine, cytarabine, and granulocyte colony stimulating factor (G-CSF) with idarubicin (FLAG-IDA), were administered during 28-day cycles.
  Interventions: Drug: Salvage Chemotherapy

INTERVENTIONS:
Drug: Quizartinib — 20 or 30 mg quizartinib tablets administered orally once daily
  Other Names: AC220
  Arms: Quizartinib
Drug: Salvage Chemotherapy — Low dose cytarabine (LoDAC); mitoxantrone, etoposide, and intermediate-dose cytarabine (MEC); or fludarabine, cytarabine, and granulocyte colony stimulating factor (G-CSF) with idarubicin (FLAG-IDA) administered during 28-day cycles
  Other Names: Standard of Care
  Arms: Salvage chemotherapy

SUMMARY:
The primary objective of the study is to determine whether quizartinib monotherapy prolongs overall survival (OS) compared to salvage chemotherapy in subjects with FMS-like tyrosine kinase 3 - Internal Tandem Duplication (FLT3-ITD) positive AML who are refractory to or have relapsed within 6 months, after first-line AML therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent approved by the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) with privacy language in accordance with national regulations (e.g., Health Insurance Portability and Accountability Act [HIPAA] authorization for United States [US] sites) prior to any study related procedures, including withdrawal of prohibited medications if applicable.
2. Age ≥ 18 years or the minimum legal adult age (whichever is greater) at the time of Informed consent.
3. Morphologically documented primary Acute Myeloid Leukemia (AML) or AML secondary to Myelodysplastic Syndrome (MDS), as defined by World Health Organization (WHO) criteria, as determined by pathology review at the study site.
4. In first relapse (with duration of remission of 6 months or less) or refractory after prior therapy, with or without HSCT. Induction therapy must have included at least 1 cycle of an anthracycline/mitoxantrone-containing induction block at a standard dose.
5. Presence of the FLT3-ITD activating mutation in bone marrow or peripheral blood (allelic ratio as determined by a central laboratory with a cutoff of ≥3% FLT3-ITD/total FLT3). If a specimen has been sent for FLT3-ITD testing at the central laboratory but the subject requires treatment for AML before the central FLT3-ITD test result is available, a local test result may be acceptable for randomization after consultation with the Medical Monitor.
6. Eligibility for pre-selected salvage chemotherapy, according to the Investigator's assessment.
7. Eastern Cooperative Oncology Group (ECOG) performance score 0-2.
8. Discontinuation of prior AML treatment before the start of study treatment (except hydroxyurea or other treatment to control leukocytosis) for at least 2 weeks for cytotoxic agents, or for at least 5 half-lives for non cytotoxic agents.
9. Serum creatinine ≤1.5×upper limit of normal (ULN), or glomerular filtration rate >25 mL/min, as calculated with the Cockcroft-Gault formula.
10. Serum potassium, magnesium, and calcium (serum calcium corrected for hypoalbuminemia) within institutional normal limits. Subjects with electrolytes outside the normal range will be eligible if these values are corrected upon retesting following any necessary supplementation.
11. Total serum bilirubin ≤1.5×ULN.
12. Serum aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤2.5×ULN.

Exclusion Criteria:

1. Acute Promyelocytic Leukemia (AML subtype M3).
2. AML secondary to prior chemotherapy for other neoplasms, except AML secondary to prior Myelodysplastic Syndrome (MDS).
3. History of another malignancy, unless the candidate has been disease-free for at least 5 years.
4. Persistent, clinically significant > Grade 1 non-hematologic toxicity from prior AML therapy.
5. Clinically significant graft versus host disease (GVHD) or GVHD requiring initiation of treatment or treatment escalation within 21 days, and/or > Grade 1 persistent or clinically significant non hematologic toxicity related to HSCT.
6. History of or current, central nervous system involvement with AML.
7. Clinically significant coagulation abnormality, such as disseminated intravascular coagulation.
8. Prior treatment with quizartinib or participated in a prior quizartinib study.
9. Prior treatment with a FLT3 targeted therapy including sorafenib or investigational FLT3 inhibitors (not including the multi-kinase inhibitor, midostaurin).
10. Major surgery within 4 weeks prior to screening.
11. Radiation therapy within 4 weeks prior to screening.
12. Uncontrolled or significant cardiovascular disease
13. Active infection not well controlled by antibacterial or antiviral therapy.
14. Known infection with human immunodeficiency virus, or active hepatitis B or C, or other active clinically relevant liver disease.
15. Unwillingness to receive infusion of blood products according to the protocol.
16. In a man whose sexual partner is a woman of childbearing potential, unwillingness or inability of the man or woman to use a highly effective contraceptive method for the entire study treatment period for at least 3 months after study completion. Male subjects must not freeze or donate sperm starting at Screening and throughout the study period, and 105 days after the final study drug administration.
17. In a heterosexually active woman of childbearing potential, unwillingness or inability to use a highly effective contraceptive method for the entire study treatment period and for at least 3 months after study treatment completion. Additionally, for women randomized to chemotherapy, unwillingness to adhere to the restrictions in the respective locally established guidelines and local approved label (prescribing information, Summary of Product Characteristics, or US product insert) from the manufacturer and the Patient Information Leaflet (package insert) as instructed by the Investigator.
18. Pregnancy.
19. Female Subjects must agree to not breastfeed from the time of Screening and throughout the study period, and for 25 days after the final study drug administration.
20. Medical condition, serious intercurrent illness, or other circumstance that, in the Investigator's judgment, could jeopardize the candidate's safety as a study subject, or that could interfere with study objectives.
21. For subjects in the United Kingdom only: Refusal of permission to allow the subject's General Practitioner to be notified of their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2020-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E. Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center; Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (131):
- United States (36):
  - City of Hope National Medical Center, Duarte, California
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - UC Davis Cancer Center, Sacramento, California
  - Stanford University Medical Center Stanford Comprehensive Cancer Center, Stanford, California
  - Yale University, New Haven, Connecticut
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Franciscan Alliance, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute Inc, Westwood, Kansas
  - LSU Health Sciences Center Feist Weiller Cancer Center, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - NY Medical College, Valhalla, New York
  - UNC Linebreger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke Cancer Institute at Duke University Health System, Durham, North Carolina
  - Wake Forest University Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health and Science University Knight Cancer Institute, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Center, The University of Texas, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Australia (6):
  - The Canbera Hospital, Garran, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Alfred Hospital, Melbourne, Victoria
- Belgium (3):
  - ZNA Stuivenberg, Antwerp, BE
  - UCL St Luc, Brussels, BE
  - Leuven UZ Gasthuisberg, Leuven, BE
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Princess Margaret Cancer Centre Princess Margaret Hospital, Toronto, Ontario
- Croatia (2):
  - Klinička Bolinca Merkur, Zagreb
  - Kliničko Bolnički Centar Zagreb, Zagreb
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
- France (10):
  - CHU de Caen, Caen
  - Centre Hospitalier Universitaire Grenoble Hopital Michalon, Grenoble
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hopital de la Conception, Marseille
  - Centre Hospitalier Universitaire Nantes, Nantes
  - Hôpital Saint Louis, Paris
  - Hopital Saint-Antoine, Paris
  - Hopital Haut Leveque Centre Francois Magendie, Pessac
  - Centre Henri-Becquerel, Rouen
  - Centre Hospitalier Universitaire Purpan, Toulouse
- Germany (14):
  - Charité Universitätsmedizin Berlin, Berlin
  - Charité Campus Virchow Klinikum, Berlin
  - Klinikum Braunschweig, Braunschweig
  - Universitatsklinikum Dresden, Dresden
  - Klinikum der Johann Wolfgang-Goethe-Universität, Frankfurt
  - Universitätsklinikum Halle, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Uniklinik Heidelberg Medizinische Klinik und Poliklinik V, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - University Mainz, Mainz
  - Universitätsklinikum Giessen und Marburg GmbH, Marburg
  - LMU München Klinikum Großhadern, München
  - Medizinische Klinik A Hämatologie Hämostaseologie Internistische Onkologie und Pneumologie, Münster
- Hong Kong (2):
  - The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong
  - The University of Hong Kong, Queen Mary Hospital, Hong Kong
- Hungary (3):
  - Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar Szent Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont, Belgyogyaszati Intezet, Debrecen, Hajdú-Bihar
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar I. Belgyogyaszati Klinika, Budapest, Pest County
- Italy (14):
  - AOU Policlinico Consorziale di Bari, Bari
  - Università di Bologna, Bologna
  - Unità Operativa di Ematologia e Unità Operativa CTMO, Cagliari
  - Arcispedale S Anna, Ferrara
  - AOU Careggi, Florence
  - IRCCS Azienda Ospedaliera Universitaria San Martino, Genova
  - Opsedale San Martino di Genova, Genova
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliero Universitaria San Luigi Gonzaga, Orbassano
  - L'UOC di Ematologia del Policlinico Tor Vergata, Rome
  - Policlinico Universitario Agostino Gemelli, Rome
  - Azienda Ospedaliero Universitaria Senese, Policlinico S. Maria alle Scotte, Siena
  - Ospedale di Circolo-a Fondazione Macchi, Varese
- Netherlands (3):
  - VU Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
- Poland (3):
  - Uniwersytecki Szpital Kliniczny w Biatymstoku, Klinika Hematologii z Pododzialem Chorob Naczyn, Bialystok
  - Samodzielny Publiczny Szpital Kliniczny im. Andrzeja Mieleckiego Slaskiego Uniwersytetu Medycznego w Katowicach Oddzial Hematologii i Transplantacji Szpiku, Katowice
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Klinika Hematoonkologii i Transplantacji Szpiku, Lublin
- Serbia (2):
  - Klinicki Centar Srbije, Belgrade
  - Klinicki Centar Vojvodine, Novi Sad
- Singapore (2):
  - National University of Singapore, Singapore
  - Singapore General Hospital, Singapore
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (8):
  - Hospital Son Espases, Palma, De Mallorca
  - Hospital La Fe, Valencia, SP
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (7):
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Saint James University Hospital, Leeds, England
  - King's College Hospital, London, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Royal Marsden Hospital Sutton, Sutton, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - University Hospital of Wales, Cardiff, South Glamorgan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Kang D, Ludwig E, Jaworowicz D, Huang H, Fiedler-Kelly J, Cortes J, Ganguly S, Khaled S, Kramer A, Levis M, Martinelli G, Perl A, Russell N, Abutarif M, Choi Y, Yin O. Concentration-QTc analysis of quizartinib in patients with relapsed/refractory acute myeloid leukemia. Cancer Chemother Pharmacol. 2021 Apr;87(4):513-523. doi: 10.1007/s00280-020-04204-y. Epub 2021 Jan 8. PMID 33415416
- [Derived] Cortes JE, Khaled S, Martinelli G, Perl AE, Ganguly S, Russell N, Kramer A, Dombret H, Hogge D, Jonas BA, Leung AY, Mehta P, Montesinos P, Radsak M, Sica S, Arunachalam M, Holmes M, Kobayashi K, Namuyinga R, Ge N, Yver A, Zhang Y, Levis MJ. Quizartinib versus salvage chemotherapy in relapsed or refractory FLT3-ITD acute myeloid leukaemia (QuANTUM-R): a multicentre, randomised, controlled, open-label, phase 3 trial. Lancet Oncol. 2019 Jul;20(7):984-997. doi: 10.1016/S1470-2045(19)30150-0. Epub 2019 Jun 4. PMID 31175001
- [Derived] Cortes J, Perl AE, Dohner H, Kantarjian H, Martinelli G, Kovacsovics T, Rousselot P, Steffen B, Dombret H, Estey E, Strickland S, Altman JK, Baldus CD, Burnett A, Kramer A, Russell N, Shah NP, Smith CC, Wang ES, Ifrah N, Gammon G, Trone D, Lazzaretto D, Levis M. Quizartinib, an FLT3 inhibitor, as monotherapy in patients with relapsed or refractory acute myeloid leukaemia: an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2018 Jul;19(7):889-903. doi: 10.1016/S1470-2045(18)30240-7. Epub 2018 May 31. PMID 29859851

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 367 participants who met the inclusion and none of the exclusion criteria were randomized (intent-to-treat population); 335 received study drug (safety analysis set).
Pre-assignment Details: Prior to randomization, the investigator was required to pre-select 1 of the 3 salvage chemotherapy regimens for each participant. Randomization was stratified by response to prior therapy (relapsed in ≤6 months [with or without HSCT] or refractory) and pre-selected salvage chemotherapy (high or low intensity chemotherapy) for all participants.
Period: Overall Study
Arm/Group | Quizartinib | Salvage Chemotherapy
Started | 245 | 122
Ongoing (as of Data Cutoff) | 45 | 16
Did Not Receive Treatment | 4 | 28
Completed | 200 | 106
Not Completed | 45 | 16

BASELINE CHARACTERISTICS:
Population: Participants received standard of care salvage chemotherapy (administered subcutaneously [LoDac] or intravenously [MEC and FLAG-IDA]).
Groups:
- Total: Total of all reporting groups
Arm/Group | Quizartinib | Salvage Chemotherapy | Total
Number analyzed (Participants) | 245 | 122 | 367
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 180 | 89 | 269
  >=65 years | 65 | 33 | 98
Age, Continuous [Median (Full Range); unit: years] | 55.0 [19 to 81] | 57.5 [18 to 78] | 56.0 [18 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 58 | 190
  Male | 113 | 64 | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 24 | 16 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 3 | 12
  White | 184 | 93 | 277
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 27 | 10 | 37
Region of Enrollment [Number; unit: participants]
  Singapore | 0 | 2 | 2
  Hong Kong | 5 | 3 | 8
  Hungary | 1 | 0 | 1
  United States | 82 | 36 | 118
  Czechia | 2 | 0 | 2
  United Kingdom | 21 | 14 | 35
  Spain | 15 | 6 | 21
  Canada | 18 | 5 | 23
  Netherlands | 2 | 1 | 3
  South Korea | 11 | 7 | 18
  Belgium | 1 | 0 | 1
  Taiwan | 2 | 1 | 3
  Poland | 2 | 0 | 2
  Italy | 34 | 19 | 53
  Australia | 3 | 3 | 6
  France | 20 | 7 | 27
  Serbia | 1 | 0 | 1
  Germany | 25 | 18 | 43

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in Participants That Received Quizartinib Versus Salvage Chemotherapy
Description: Overall Survival is defined as the time (in weeks) from the date of randomization to the date of death due to any cause. Median and quartiles are calculated using the Kaplan-Meier method.
Time Frame: At approximately 3 years 9 months
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Quizartinib | Salvage Chemotherapy
Number analyzed (Participants) | 245 | 122
weeks | 27.0 [15.4 to 62.6] | 20.4 [8.3 to 39.6]
Statistical Analysis 1: Comparison: Quizartinib vs Salvage Chemotherapy; Stratified analysis - stratification factors include prior therapy and response (Relapsed in ≤6 months (not post-HSCT), Refractory, or relapsed in ≤6 months post allogeneic HSCT), and pre-selected chemotherapy (High intensity chemotherapy [MEC or FLAG-IDA], or low intensity chemotherapy [LoDAC]); Test type: Other; p = 0.0185, P-value for HR=1 (1-sided); Hazard Ratio (HR) = 0.758, 95% CI 2-sided [0.584 to 0.983]

2. Secondary Outcome: Event-free Survival in Participants That Received Quizartinib Versus Salvage Chemotherapy
Description: Event-free survival is defined as the time (in weeks) from randomization until documented refractory disease, relapse after complete composite remission (CRc), or death from any cause, whichever is observed first.
Time Frame: At approximately 3 years 9 months
Population: Event-free survival was assessed in the intent-to-treat (ITT) analysis set.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Quizartinib | Salvage Chemotherapy
Number analyzed (Participants) | 245 | 122
weeks | 6.0 [0.1 to 19.7] | 3.7 [0.1 to 17.0]
Statistical Analysis 1: Comparison: Quizartinib vs Salvage Chemotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2034, P value for HR=1 (1-sided); Hazard Ratio (HR) = 0.898, 95% CI 2-sided [0.697 to 1.157]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the first dose of study drug to 30 days after the last dose (or longer if assessed as treatment related). All safety events are reported for participants in the Safety Analysis Set who received at least 1 dose of study drug or salvage chemotherapy.
Description: Differences in treatment regimens make the Treatment-emergent adverse events (TEAE) collection period span multiple 28-day cycles in the Quizartinib arm and only 1-2 weeks in the salvage chemotherapy arm.
Arm/Group | Quizartinib | Salvage Chemotherapy
All-Cause Mortality (participants affected / at risk) | 80/241 | 16/94
Serious Adverse Events (participants affected / at risk) | 168/241 | 37/94
Other Adverse Events (participants affected / at risk) | 238/241 | 91/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quizartinib (N=241) | Salvage Chemotherapy (N=94)
Phlebitis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Graft versus host disease in intestine (Immune system disorders) | 4 | 0
Graft versus host disease in liver (Immune system disorders) | 1 | 0
Graft versus host disease in skin (Immune system disorders) | 3 | 0
Chills (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Edema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 8 | 2
Vascular complication associated with device (General disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural hematoma (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural hemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 5 | 0
Liver function test abnormal (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 2 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 50 | 9
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Cerebral hemorrhage (Nervous system disorders) | 2 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Hemorrhage intracranial (Nervous system disorders) | 5 | 2
Headache (Nervous system disorders) | 1 | 0
Horner's syndrome (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 5 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Melena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0
Hematuria (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalized (Skin and subcutaneous tissue disorders) | 2 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Acarodermatitis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Anal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 4 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 6 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 3 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0
Enterobacter bacteremia (Infections and infestations) | 1 | 0
Enterobacter infection (Infections and infestations) | 3 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Escherichia bacteremia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 2 | 3
Fungal skin infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 3 | 0
Lymph gland infection (Infections and infestations) | 1 | 0
Necrotizing fascitis (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 2 | 0
Neutropenic sepsis (Infections and infestations) | 7 | 2
Peritonitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 22 | 3
Pneumonia fungal (Infections and infestations) | 3 | 2
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Pulmonary mycosis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 16 | 4
Septic shock (Infections and infestations) | 5 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 2 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal bacteremia (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 4 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Stenotrophomonas infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 0
Urinary tract infection (Infections and infestations) | 6 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulval cellulitis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quizartinib (N=241) | Salvage Chemotherapy (N=94)
Hypertension (Vascular disorders) | 9 (9) | 8 (8)
Hypotension (Vascular disorders) | 32 (39) | 10 (10)
Graft versus host disease (Immune system disorders) | 14 (14) | 0 (0)
Graft versus host disease in skin (Immune system disorders) | 16 (18) | 0 (0)
Asthenia (General disorders) | 34 (38) | 10 (11)
Chills (General disorders) | 15 (15) | 7 (8)
Fatigue (General disorders) | 67 (81) | 18 (22)
Edema peripheral (General disorders) | 51 (58) | 22 (26)
Pain (General disorders) | 19 (21) | 8 (8)
Pyrexia (General disorders) | 88 (130) | 42 (69)
Anxiety (Psychiatric disorders) | 19 (21) | 4 (4)
Confusional state (Psychiatric disorders) | 7 (7) | 5 (5)
Insomnia (Psychiatric disorders) | 22 (24) | 13 (13)
Contusion (Injury, poisoning and procedural complications) | 15 (17) | 2 (2)
Alanine aminotransferase increased (Investigations) | 32 (46) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 26 (41) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 18 (24) | 4 (5)
Blood bilirubin increased (Investigations) | 24 (30) | 3 (6)
Blood creatinine increased (Investigations) | 16 (22) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 63 (90) | 2 (2)
Neutrophil count decreased (Investigations) | 31 (46) | 14 (21)
Platelet count decreased (Investigations) | 33 (39) | 12 (20)
Weight decreased (Investigations) | 27 (31) | 5 (5)
White blood cell count decreased (Investigations) | 35 (45) | 14 (17)
Sinus tachycardia (Cardiac disorders) | 8 (8) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 56 (64) | 13 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 48 (61) | 8 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 28 (34) | 8 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 (26) | 6 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 86 (131) | 29 (35)
Febrile neutropenia (Blood and lymphatic system disorders) | 41 (47) | 19 (28)
Leukocytosis (Blood and lymphatic system disorders) | 14 (14) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 13 (17) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 48 (77) | 11 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 62 (84) | 20 (21)
Dizziness (Nervous system disorders) | 36 (41) | 10 (10)
Dysgeusia (Nervous system disorders) | 22 (22) | 1 (1)
Headache (Nervous system disorders) | 51 (64) | 16 (19)
Dry eye (Eye disorders) | 13 (13) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 11 (13) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 30 (33) | 15 (16)
Abdominal pain upper (Gastrointestinal disorders) | 18 (21) | 0 (0)
Constipation (Gastrointestinal disorders) | 47 (54) | 22 (29)
Diarrhea (Gastrointestinal disorders) | 68 (98) | 34 (42)
Dry mouth (Gastrointestinal disorders) | 13 (14) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 20 (20) | 6 (6)
Gingival bleeding (Gastrointestinal disorders) | 16 (16) | 3 (3)
Nausea (Gastrointestinal disorders) | 114 (164) | 39 (47)
Proctalgia (Gastrointestinal disorders) | 8 (9) | 5 (5)
Stomatitis (Gastrointestinal disorders) | 39 (39) | 18 (18)
Vomiting (Gastrointestinal disorders) | 80 (116) | 20 (25)
Dysuria (Renal and urinary disorders) | 15 (16) | 39 (39)
Petechiae (Skin and subcutaneous tissue disorders) | 27 (31) | 6 (8)
Pruritis (Skin and subcutaneous tissue disorders) | 15 (15) | 6 (8)
Rash (Skin and subcutaneous tissue disorders) | 36 (41) | 9 (10)
Skin lesion (Skin and subcutaneous tissue disorders) | 14 (14) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (24) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (29) | 9 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 (22) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 19 (20) | 6 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (16) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (26) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 48 (62) | 10 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (17) | 7 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 (33) | 7 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 27 (36) | 10 (10)
Hypokalemia (Metabolism and nutrition disorders) | 76 (124) | 25 (45)
Hypomagnesemia (Metabolism and nutrition disorders) | 36 (56) | 7 (12)
Hyponatremia (Metabolism and nutrition disorders) | 21 (36) | 6 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 23 (31) | 10 (12)
Bacteremia (Infections and infestations) | 2 (2) | 5 (5)
Device related infection (Infections and infestations) | 9 (9) | 7 (7)
Enterococcal infection (Infections and infestations) | 1 (1) | 5 (5)
Pneumonia (Infections and infestations) | 11 (11) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 17 (17) | 1 (1)
Urinary tract infection (Infections and infestations) | 18 (26) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT02039726/Prot_SAP_000.pdf